CLINICAL TRIAL: NCT05771935
Title: Ultrasound Guided Ulnar Versus Radial Artery Cannulation in Pediatrics Undergoing Major Non Cardiac Surgery: Double Blinded Randomized Controlled Study
Brief Title: Ultrasound Guided Ulnar Versus Radial Artery in Pediatrics Undergoing Major Non Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Khaled Abdelfattah Abdallah Sarhan, principal investigator,Lecturer of anesthesia, Cairo university, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS-225-2022
Record Dates: First submitted 2023-03-05; First posted 2023-03-16 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Anesthesia; Pediatrics; Radial Artery; Ulnar Artery
Keywords: ultrasound; arterial cannulation; radial; ulnar; surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Group R) (Experimental): receive radial artery cannulation using ultrasound
  Interventions: Procedure: ultrasound guided radial versus ulnar artery cannulation
- (Group U) (Active Comparator): receive ulnar artery cannulation using ultrasound
  Interventions: Procedure: ultrasound guided radial versus ulnar artery cannulation

INTERVENTIONS:
Procedure: ultrasound guided radial versus ulnar artery cannulation — Ultrasound examination will be performed using a hockey stick, high frequency (5-10 MHz) ultrasound probe (S-NerveTM; SonoSite Inc., Bothell, WA, USA).
  . Arterial cannulation will be performed using the long axis view (in-plane) technique with a 24 or 22-gauge canulae according to the operator preference. Cannulation will be considered complete when the arterial waveform is confirmed on the monitor. If cannulation is unsuccessful within the third attempt or within 10 min, the case will be considered a failure at the chosen artery. After the failure, an alternative site will be used for cannulation and the case will be excluded from the study.

SUMMARY:
This study aims to assess the safety and efficacy of ulnar artery cannulation compared to radial artery cannulation in pediatrics undergoing major non cardiac procedures.

DETAILED DESCRIPTION:
The study is a double blinded randomized controlled trial that will be conducted at Abu Al Reesh Children's Hospital, Faculty of Medicine, Cairo University after approval of research and ethics committees.

Children will be recruited into the trial during pre-operative assessment. will be randomly assigned to one of two groups Recruited patients will be randomly allocated by a computer-generated sequence of codes using randomization software (https://www. randomizer.org) into one of the two groups; in a 1:1 ratio (Group R) to receive radial artery cannulation and (Group U) to receive ulnar artery cannulation using ultrasound. The randomization sequence will be concealed in sequentially numbered, sealed opaque envelopes. The sealed envelopes will be opened by an anesthesia nurse immediately before induction of anesthesia.

After induction of anesthesia, modified Allen's test will be done by the ultrasound operator as following:

An Esmarch bandage will be used to exsanguinate the selected hand for cannulation according to the operator preference for 30 seconds, then the operator will apply simultaneous pressure to the ulnar and radial arteries of the chosen limb to occlude them. The bandage will then be released. Next, the pressure over the opposed artery selected for cannulation will be released and the time (in seconds) it takes for color to return to the hand will be measured.

Allen test results will be interpreted as follows:

If color returns to the hand within 5 seconds, the result of the Allen test is negative (normal) and the artery can safely be cannulated.

If color does not return to the palm within 5 seconds, the test result is positive (abnormal). The test will be repeated on the other hand and if the test is positive another site will be selected for cannulation, and the patient will be excluded from the study.

The patient's wrist will be extended over a roll to keep the angle of the wrist unchanged to 30- 45 degrees. After hand washing and sterile gloving; skin will be prepared using alcohol-based chlorhexidine antiseptic in both groups.

Assessment of proposed artery for cannulation using ultrasonography will be performed by one of 2 pediatric anesthesiologists blinded to group allocation who have performed more than 50 ultrasound guided arterial cannulation in pediatrics.

Ultrasound examination will be performed using a hockey stick, high frequency (5-10 MHz) ultrasound probe (S-NerveTM; SonoSite Inc., Bothell, WA, USA).

Image depth will be set to 2- 3 cm and gain settings adjusted to enhance views. Both external force and the angle will be manipulated to optimize images.

The radial artery will be identified in the transverse plane and confirmed with color flow doppler, then in the longitudinal plane by rotating the probe 90 degrees clockwise while maintaining the arterial image. This method will be repeated for the ulnar artery. All antro-posterior (AP) and transverse (T) diameters will be made at the inner (intimal) edge of the vessel. AP diameter will be measured on both transverse and longitudinal images. Cross-sectional area (CSA) will be calculated then as following: π [AP × T] /4. Three measurements will be collected, and the average values will be used for analysis.

Arterial cannulation will be performed using the long axis view (in-plane) technique with a 24 or 22-gauge canulae (Euromed For Medical Industries, S.A.E., Cairo, Egypt) according to the operator preference. Cannulation will be considered complete when the arterial waveform is confirmed on the monitor. If cannulation is unsuccessful within the third attempt or within 10 min, the case will be considered a failure at the chosen artery. After the failure, an alternative site will be used for cannulation and the case will be excluded from the study. The overall procedure time of arterial cannulation is defined as the time interval from the first skin puncture by the canula to confirmation of the arterial waveform on the monitor. After the procedure, the diameter of the cannulated artery and the occurrence of hematoma or vasospasm will be evaluated with ultrasound. Data will be collected by another anesthesiologist who is blinded to the group allocation.

ELIGIBILITY:
Inclusion Criteria:

- All pediatrics ASA I&II aged 1 month -10 years undergoing major non cardiac surgeries.

Exclusion Criteria:

* • Patients undergoing cardiac surgeries.

  * Refusal of parents.
  * Ischemia defined as (color changes: blanching, duskiness, and or change in temperature of the extremity used for cannulation compared to the contralateral one).
  * Previous arterial cannulation within last week.
  * Patients requiring inotropic support before the start of procedures.
  * Rash or signs of infection or hematoma at the site of cannulation.
  * Patients requiring emergency procedures.

Ages: 1 Month to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2023-03-05 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Rate of successful cannulation at first attempt | 15 minutes
  (the procedure will be classified as successful when the artery is cannulated, and an arterial waveform is recorded within less than 3 attempts and or 15 minutes from the first puncture).

SECONDARY OUTCOMES:
diameters of the arteries before cannulation | preoperative
  Anteroposterior, transverse diameters and cross-sectional area of the arteries before cannulation
diameters of the arteries after cannulation | 15 minutes from start of cannulation
  Anteroposterior, transverse diameters and cross-sectional area of the arteries after cannulation
incidence of vasospasm | 15 minutes from start of cannulation
  more than 25% decrease in the artery diameter after cannulation without intra-arterial hematoma.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university hospitals, kasralainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided